CLINICAL TRIAL: NCT06597474
Title: Food-Body-Mind Intervention: Promote Whole Child Health
Brief Title: Food-Body-Mind Intervention (16 Weeks)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Jiying Ling, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00009256-MOD00007491
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Wellness; Emotional Problem; Behavioral Problem of Child; Social Skills; Obesity, Childhood
Keywords: Mindfulness; Mindful eating; Yoga; Deep breathing; Family; Prevention
MeSH Terms: conditions — Social Skills; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Two-group cluster RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food-Body-Mind intervention (Experimental): Guided by the Actor-Partner Interdependence Model, the Allostatic Load Model, and the Transactional Theory of Stress and Coping, the proposed 16-week Food-Body-Mind intervention includes: 1) a school-based mindfulness component delivered to equip preschoolers with knowledge and skills in mindful eating and movement (e.g., yoga, deep breathing exercises); 2) a home-based mindfulness component to increase caregivers' skills in practicing mindful eating, movement, and parenting behaviors at home to foster a more positive, mindful, and healthy home environment; and 3) a school learning and home practice connection component to improve caregiver-preschooler relationships.
  Interventions: Behavioral: Food-Body-Mind
- Usual care control (No Intervention): Like those in the intervention group, preschoolers assigned to the control group will receive usual Head Start activities during the intervention period. After the 12-month follow-up data collection from both intervention and control participants in each year, each control family will receive all intervention supplies including the "Tasty Healthy Cookbook," "MyPlate" plates, and a breathing ball, as well as the program manual on how to use the intervention supplies. These intervention supplies will be distributed to control families at the end of in-person data collection appointments. Moreover, a virtual caregiver meeting on mindful eating, movement, and parenting will be provided to all caregivers who are interested.

INTERVENTIONS:
Behavioral: Food-Body-Mind — The Food-Body-Mind intervention includes 3 main components: 1) a school-based mindfulness component delivered by daycare teachers to equip preschoolers with knowledge and skills in mindful eating and movement (e.g., yoga, deep breathing exercises) to reduce emotional eating and increase F/V intake and physical activity; 2) a home-based mindfulness component to increase caregivers' skills in practicing mindful eating, movement, and parenting behaviors at home to foster a more positive, mindful, and healthy home environment; and 3) a preschooler school learning and caregiver home practice connection component to improve caregiver-preschooler relationships.
  Arms: Food-Body-Mind intervention

SUMMARY:
This novel, timely, and theory-driven Food-Body-Mind intervention addresses the national emergency of mental health crises in early childhood. By targeting Head Start racially/ethnically diverse preschoolers from low-income backgrounds in both urban and rural areas, this intervention is expected to contribute toward reducing health disparities and promoting health equity, a major priority of the NIH and Healthy People 2030. If effective, it can be scalable to Head Start programs across urban and rural settings nationally with long-term sustainability benefits.

DETAILED DESCRIPTION:
Mental, emotional, and behavioral (MEB) disorders begin in early childhood, with one in six US preschoolers aged 3-5 years diagnosed with a MEB disorder. Children from low income and economically marginalized (LIEM) backgrounds have a higher risk of being diagnosed with MEB disorders than those from higher income families. To address the mental and physical health disparities based on socioeconomic status, ethnicity/race, and urban/rural residency, the proposed study will target Head Start racially/ethnically diverse preschoolers from LIEM backgrounds in both urban and rural areas. Guided by the Actor-Partner Interdependence Model, the Allostatic Load Model, and the Transactional Theory of Stress and Coping, the proposed 16-week Food-Body-Mind intervention includes: 1) a school-based mindfulness component delivered to equip preschoolers with knowledge and skills in mindful eating and movement (e.g., yoga, deep breathing exercises); 2) a home-based mindfulness component to increase caregivers' skills in practicing mindful eating, movement, and parenting behaviors at home to foster a more positive, mindful, and healthy home environment; and 3) a school learning and home practice connection component to improve caregiver-preschooler relationships. The purpose of this 5-year cluster randomized controlled trial is to evaluate the effects of the 16-week school- and home-based, multi-component, Food-Body-Mind intervention on improving both preschoolers' and caregivers' MEB and physical health. The long-term goal is to achieve optimal whole child health in early childhood to foster a healthier generation in the US. Fifty Head Start daycare centers will be randomized into the intervention (n=25: 8 urban and 17 rural daycare centers) or usual care control group (n=25: 8 urban and 17 rural daycare centers). Five caregiver-preschooler dyads will be recruited from each daycare classroom (total 400 dyads from 80 daycare classrooms: 200 urban dyads and 200 rural dyads). Analyses will be based on the intention-to-treat principle. The three aims are to: 1) determine effects of the intervention on improving preschoolers' mental (chronic stress by hair cortisol), emotional (sadness, fear, anger, positive affect), behavioral (problem behaviors, social skills), and physical health (BMI z-score, % body fat) from baseline (0 month) to 4 months (immediate post-intervention) and to 16 months post-baseline (12-month F/U) when compared to control group in geographically diverse urban and rural Head Start daycare sites; 2) examine intervention effects on improving caregivers' physical (BMI, % body fat, blood pressure) and mental (stress, anxiety, depression) health from 0 to 4 months and to 16 months (12-month F/U) compared to control; and 3) explore the potential mediators (caregiver mindfulness, physical activity, F/V intake, caregiver-preschooler relationship, and caregiver coping) of intervention effects on preschoolers' MEB and physical health and caregivers' physical and mental health from 0 to 4 months and to 16 months (12-month F/U). Results from this study will improve the evidence base of complementary and integrative health approaches that can be delivered in geographically diverse daycare settings.

ELIGIBILITY:
Inclusion Criteria:

1. Parental consent and child (if the child is 5 years) verbal assent received
2. Children are 3-5 years old attending a Head Start program and caregivers are the primary adult caregivers for the children
3. Caregivers are willing to use Facebook or the private program website for participation
4. Participants have at least weekly internet access using a smartphone, a tablet, or a computer

Exclusion Criteria:

1. preschoolers who have a motor disability or impairment (e.g., cerebral palsy, spinal cord injury, lost or damaged limb, motor skills disorder, muscular dystrophy, spina bifida) preventing them from participating in any physical activity;
2. preschoolers who have a diagnosed medical condition (e.g., phenylketonuria, pediatric malabsorption syndrome, pollen food allergy syndrome) requiring a restrict diet and precluding them from any dietary changes particularly fruit/vegetable intake; and
3. preschoolers who have diagnosed disorders (e.g., autism spectrum disorder level 3) causing severe difficulty (e.g., nonverbal, cannot initiate social interaction) with communication and interaction with other people.

There will be no exclusion criterion for primary adult caregivers, as the primary focus is preschoolers and caregivers serve as a support role.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Preschoolers' problem behaviors | Change from Month 0 (Time 1) to Month 4 (Time 2)
  Problem behaviors will be assessed by the Preschool and Kindergarten Behavior Scales-Second Edition (PKBS-2). The Problem Behavior scale includes 42 items on 2 subscales: Externalizing Problems and Internalizing Problems. Total standard scores (M=100, SD=15) will be calculated, with a higher score indicating a higher level of problem behaviors. Preschoolers' problem behaviors rated by teachers will be the primary outcome, and problem behaviors rated by caregivers will be the secondary outcome.

SECONDARY OUTCOMES:
Preschoolers' problem behaviors | Change from Month 4 (Time 2) to Month 16 (Time 3)
  Problem behaviors will be assessed by the Preschool and Kindergarten Behavior Scales-Second Edition (PKBS-2). The Problem Behavior scale includes 42 items on 2 subscales: Externalizing Problems and Internalizing Problems. Total standard scores (M=100, SD=15) will be calculated, with a higher score indicating a higher level of problem behaviors.
Preschoolers' social skills | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Social skills will be assessed by the Preschool and Kindergarten Behavior Scales-Second Edition (PKBS-2). The Social Skills scale includes 34 items on 3 subscales: Social Cooperation, Social Interaction, and Social Independence. Total standard scores (M=100, SD=15) will be calculated, with a higher score indicating a higher level of social skills.
Preschoolers' sadness | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Sadness will be assessed by the 7-item National Institutes of Health (NIH) Toolbox Sadness Parent Report Fixed Form. Response choices for the 3-Likert scale include: never or not true, sometimes or somewhat true, and often or very true. A total raw score was calculated and then transformed to the uncorrected T-scores (M=50, SD=10). A higher T-score indicates a higher level of sadness reported by parents/caregivers.
Preschoolers' fear | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Fear will be assessed by the 6-item, 3-Likert (never or not true, sometimes or somewhat true, often or very true) NIH Toolbox Fear-Over Anxious Parent Report Fixed Form. A total raw score was calculated and then transformed to the uncorrected T-scores (M=50, SD=10). A high T-score indicates a higher level of fear.
Preschoolers' anger | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Anger will be assessed using the 9-item, 3-Likert (never or not true, sometimes or somewhat true, often or very true) NIH Toolbox Anger Parent Report Fixed Form. A total raw score was calculated and transformed to the uncorrected T-scores (M=50, SD=10). A higher T-score indicates a higher level of child anger.
Preschoolers' positive affect | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Positive affect will be assessed by the 9-item NIH Toolbox Positive Affect Parent Report Fixed Form. Each question has five response choices: not at all, a little bit, somewhat, quite a bit, and very much. A total raw score was calculated and then transformed to the uncorrected T-scores (M=50, SD=10). A higher T-score indicates a higher level of positive affect.
Dyads' BMI | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Height will be measured to the nearest 0.1cm using the Shorr board, and weight will be measured to the nearest 0.1kg using the Seca 874 scale or the portable InBody 270 body composition analyzer. The online SAS program for Centers for Disease Control and Prevention Growth Charts was applied to calculate preschoolers' BMI for age and sex.
Dyads' percent body fat | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Percent body fat will be measured to the nearest 0.1% using the portable InBody 270 body composition analyzer (FDA cleared medical device). When measuring % body fat, each participant's study ID, biological sex, age, and height will be entered into the scale. After the setup, each participant will be instructed to step on the scale surface and align feet with the food electrodes. When prompted, each participant will grab the hand electrodes by placing their thumbs on the thumb electrodes and wrapping their fingers around the bottom electrodes.
Preschoolers' chronic stress | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Preschoolers' chronic stress will be assessed by hair cortisol concentration level. A proximal 3-cm segment hair sample, weighing approximately 20 mg, will be cut from 2-3 locations at the posterior vertex of each preschooler's head with a stainless-steel styling shear. Hair samples (labeled at the root ends furthest away from the head) will be stored in an aluminum foil pouch at room temperature. The hair samples will be analyzed by the Child Study Center lab at the Yale University. Cortisol in pg/mg will be extracted from the powdered hair by incubation with methanol for 18-24 hours.
Dyads' physical activity | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Actigraph (wGT3X-BT; 7-day period) worn on hip by both preschoolers and caregivers will be used to measure physical activity. Before distributing the ActiGraph to dyads for wearing, investigators will use the ActiLife software to initialize each ActiGraph and set to begin data collection at 5 AM on the day after dyads receive the ActiGraph from data collectors. When distributing the ActiGraph to dyads, the "superhero with a magic belt" story will be shared with preschoolers to encourage them to wear the ActiGraph for 7 consecutive days, and written wear instructions will be provided to caregivers: right hip (attached to belt) from time getting out of bed in AM to going to sleep at night for 7 consecutive days (not worn bathing/swimming).
Dyads' fruit/vegetable intake | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Fruit/vegetable intake will be assessed by the skin carotenoid levels via Veggie Meter® as well as a 2-question survey. Each participant's non-dominant index finger will be used, and the average of three scans with a range of 0-850 will be recorded as the final score. A high Veggie Meter score indicates a higher level of fruit/vegetable intake. For the 2-question survey, a sum score with a range of 0-10 will be calculated, with a higher score indicating a higher level of fruit/vegetable intake.
Caregivers' blood pressure | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Systolic and diastolic blood pressure will be assessed by the SunTech CT40 device. Investigators will follow the procedures in the Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: 1) Caffeine, exercise, and smoking will be avoided for at least 30 minutes before measurement; 2) The caregiver will be seated quietly for at least 5 minutes in a chair, with feet on the floor and arms supported at heart level; 3) An appropriate sized cuff (cuff bladder encircling at least 80% of the arm) will be used on the left arm unless having a surgery or injury; 4) Two measurements will be taken at 1 minute interval and averaged for recording; and 5) The caregiver will receive their blood pressure reading in writing as well as the American Heart Association Blood Pressure Fact Sheet demonstrating the blood pressure categories, strategies for controlling blood pressure, and blood pressure resources.
Caregiver-preschooler relationship | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Caregiver-preschooler relationship will be measured by the 15-item Child-Parent Relationship Scale - Short Form (CPRS-SF), which is a 5-point Likert scale with 2 subscales: conflict and closeness. Sum scores (range for conflict subscale is 8-40, range for closeness subscale is 8-35) will be calculated, with a higher sum score indicating a higher level of relationship.
Caregiver mindfulness | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Caregiver mindfulness will be assessed by the 15-item Mindful Attention Awareness Scale, which is a 6-point Likert scale to assess trait mindfulness. A mean score (min-max: 1-6) will be calculated, with a higher mean score indicating a higher level of mindfulness.
Caregiver coping | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Parental coping strategies (problem-focused, emotion-focused, and avoidant coping) will be measured by the 28-item Coping Orientation to Problems Experienced Inventory (Brief-COPE). It is a 4-point Likert scale. Mean scores (min-max: 1-4) will be calculated for each coping category, with a higher mean score indicating a higher level of coping.
Household food insecurity | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  The U.S. Household Food Security Survey Module will be used to assess household, parent, and preschooler food insecurity status. Raw sum score will be calculated for each outcome (household food insecurity raw score range is 0-18, raw score range for adult food insecurity is 0-10, raw score range for child food insecurity is 0-8) and then divided into food insecure and food secure categories. A higher raw score indicates a higher level of food insecurity.
Home environment | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Home environment will be assessed by the 20-item Family Nutrition and Physical Activity Screening Tool.t has two subscales: eating and physical activity home environment. A sum score, with a range of 10-80 will be calculated, with a higher sum score indicating a healthier home environment.
Caregivers' anxiety | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Caregivers' anxiety will be measured by the Patient Health Questionnaire (PHQ)-4. The PHQ-4 is a questionnaire answered on a four-point Likert-type scale. It has the two-item measure for anxiety (Generalized Anxiety Disorder, GAD-2). The total GAD-2 score (range 0-6) will be calculated, with a higher score indicating a higher level of anxiety.
Caregivers' stress | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Caregivers' stress will be assessed by the 10-item Perceived Stress Scale. It is a 5-point Likert scale, with response choices of never to very often. A sum score (range: 0-40) will be calculated, with a higher sum score indicating a higher level of perceived stress.
Caregivers' depression | Change from Month 0 (Time 1) to Month 4 (Time 2), and change from Month 4 (Time 2) to Month 16 (Time 3)
  Caregivers' depression will be measured by the Patient Health Questionnaire (PHQ)-4. The PHQ-4 is a questionnaire answered on a four-point Likert-type scale. It has the two-item measure for depression (PHQ-2). The total PHQ-2 score (range 0-6) will be calculated, with a higher score indicating a higher level of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Action Agency, Jackson, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be shared with other researchers upon request.

REFERENCES:
- [Derived] Ling J, Kao TA, Robbins LB, Wahman CL, Kerver JM, Resnicow K, Zhang N, Lalonde H, Xie Y, Baumgartner J. Food-Body-Mind study protocol: A mindfulness-based lifestyle intervention to promote whole child health among preschoolers from economically marginalized families. Contemp Clin Trials. 2026 Jan;160:108146. doi: 10.1016/j.cct.2025.108146. Epub 2025 Nov 19. PMID 41265832